CLINICAL TRIAL: NCT02679924
Title: A Single Center, Prospective, Randomized, Sham Controlled, Double Blind, Split Face Trial Using Micro-injections of Transparent Hyaluronic Acid Gel (Restylane® Silk) for Rejuvenation of the Aging Cheek
Brief Title: A Slit Face Trial Using Micro-injections of Transparent Hyaluronic Acid Gel for Rejuvenation of the Cheek
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Isabella Guiha (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor-Investigator, Isabella Guiha, Mitchel P. Goldman, MD (Principal Investigator), Goldman, Butterwick, Fitzpatrick and Groff
Organization: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RS-2015-01
Record Dates: First submitted 2015-11-11; First posted 2016-02-11 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Problem of Aging
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restylane Silk (Experimental): Micro-injections of Restylane® Silk Hyaluronic Acid filler for correction of mid to low cheek fine lines and wrinkles.
  Interventions: Device: Hyaluronic Acid filler
- Sham Comparator (Sham Comparator): Micro-injections of normal saline for correction of mid to low cheek fine lines and wrinkles.
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Device: Hyaluronic Acid filler — The objective of this study is to determine the efficacy and safety of Restylane® Silk Hyaluronic Acid filler microinjections when used in a grid-like injection pattern for the correction of fine lines to the cheeks.
  Other Names: Restylane Silk
  Arms: Restylane Silk
Other: Sham Comparator — Micro-injections of normal saline for correction of mid to low cheek fine lines and wrinkles.
  Other Names: Normal Saline
  Arms: Sham Comparator

SUMMARY:
Soft tissue augmentation with injectable hyaluronic acid (HA) is a well-established modality for the correction of facial volume loss, fat atrophy, fine lines, and wrinkles. HA is a glycosaminoglycan that is composed of repeating D-glucuronic acid and D-N-acetylglucosamine disaccharide units. Because HA is a natural and inert constituent of the dermis, it represents an ideal substance for soft tissue augmentation. Current FDA-approved HA fillers are typically utilized to either directly target specific cutaneous rhytids or to restore overall contours by placement into fat pads or along bony structures that have remodeled with age. Restylane® Silk is a transparent injectable HA gel that received FDA approval in June 2014 for use in the lips and peri-oral region. Its unique synthesis results in smaller and finer particles that demonstrate significant hygroscopic properties and give rise to the potential for unique applications. One such application concerns the concept of "skin boosting" whereby microaliquots of HA are placed into the skin to induce biophysical improvement in dermal characteristics (1). Using this technique, a recent split-body study by Streker et al. demonstrated significant aesthetic improvements in face, hands and décolletage (2). However, there have been no well-controlled studies with validated aesthetic outcomes utilizing Restylane® Silk in this fashion to date. Because of the unique combination of ultra-fine product and high water-attracting capability, the investigators hypothesize that microinjections of Restylane® Silk can be used in a grid-like injection pattern for rejuvenation of the aging cheek.

DETAILED DESCRIPTION:
This is a single center, prospective, randomized, sham-controlled, double-blind, split-face trial using micro-injections of Restylane® Silk for correction of mid to low cheek fine lines and wrinkles. Twenty (20) subjects will be enrolled. Each subject will receive Restylane® Silk to a defined area of mid to low cheek in a randomized blinded fashion with the contralateral cheek treated by sham injection. The injections will be delivered intradermally 1mm in depth via multiple 0.02 cc microinjections distributed in a grid array pattern with 0.5 cm to 1 cm between each injection point over total treatment area. The sham injections will be administered in identical fashion and will consist of sterile normal saline. Following completion of injection treatment, manual massage will be applied to the full area to promote even distribution of the product. The maximum amount of Restylane Silk to be used per treatments session/per cheek for balancing treatment is1cc (not to exceed a total of 3cc) per treated patient. Three dimensional digital photography utilizing the Vectra 3D System (Canfield) will be utilized to document pre-treatment status, sites of injection, and post-treatment effect. Subjects will be followed up at 1 week, 2 week, 4 week, day 90, and day 180 time points. At the Day 180 time point, every subject will be given the option to receive touch up and balancing treatments to both cheeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female in general good health age 18 or over.
* Mild to moderate static rhytids involving at least a 9 cm2 area of the mid to low cheeks.
* Must be willing to give and sign a HIPPA form, photo consent and informed consent form.
* Must be willing to comply with study dosing and complete the entire course of the study.
* Female patients will be either of non-childbearing potential defined as:

  1. Having no uterus
  2. No menses for at least 12 months
  3. Bilateral tubal ligation Or;

(WOCBP) women of childbearing potential must agree to use an effective method of birth control during the course of the study, such as:

1. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device
2. Intrauterine coil
3. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
4. Abstinence (If practicing abstinence must agree to use barrier method described above (3) if becomes sexually active).
5. Vasectomized partner (must agree to use barrier method described above (3) if becomes sexually active with un-vasectomized).

   * Negative urine pregnancy test results Baseline prior to study entry (if applicable)

Exclusion Criteria:

* Pregnant, planning pregnancy during the course of the study or breastfeeding
* Severe static rhytids to the mid to low cheeks
* Previous use of any form of soft tissue augmentation in the treatment area within the past 12 months
* Pre-existing medical or dermatologic condition in the treatment area that may affect the treatment or interpretation of treatment effect (at investigator discretion)
* Presence of tattoo and/or scar in the treatment area that in the investigators opinion would interfere with study assessments
* Use of oral/topical retinoids within 1 month of Baseline
* Previous use of botulinum toxins in the treatment area within the past 6 months
* Previous surgical procedure in the treatment area within the past 12 months
* Presence or evidence of any conditions that in the opinion of the investigator might impede the subject's ability to give consent or comply with protocol requirements.
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study
* History of non-compliance with clinical research protocols
* Ablative laser resurfacing to on their face within 12 months
* Non-ablative laser or light procedures to their face within the past 3 months
* Known allergy to Restylane® Silk or any of its constituents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in Wrinkling and Elastosis | month 6
  Efficacy will be determined based on the difference between blinded evaluator assessment of Fitzpatrick-Goldman Classification of Wrinkling and Degree of Elastosis Scale between Baseline and Month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — DCLA
Locations (1):
- Dermatology Cosmetic Laser Medical Associates of La JOlla, Inc., San Diego, California, United States